CLINICAL TRIAL: NCT06324656
Title: The Efficacy of Combining Platelet-rich Plasma With Crystallized Phenol in Pilonidal Sinus Disease Treatment in Children: A Double-blind Single-center Randomized Controlled Trial
Brief Title: The Efficacy of Combining Platelet-rich Plasma With Crystallized Phenol in Pilonidal Sinus Disease
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Necmi Kadıoğlu Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: PRP-PNS
Record Dates: First submitted 2024-03-10; First posted 2024-03-22 (Actual); Last update posted 2024-08-20 (Actual); Status verified 2024-08

CONDITIONS: Pilonidal Sinus
Keywords: pilonidal sinus; Children; platelet rich plasma
MeSH Terms: conditions — Pilonidal Sinus

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Crystallized phenol (Active Comparator): Crystallized phenol group: The patients will undergo to crystallized phenol application.
  Interventions: Procedure: crystallized phenol
- Crystallized phenol + platelet rich plasma (Experimental): Crystallized phenol + platelet rich plasma group. Alongside the crystallized phenol application + patients also will receive platelet rich plasma injections in the same session.
  Interventions: Procedure: crystallized phenol + platelet rich plasma application

INTERVENTIONS:
Procedure: crystallized phenol + platelet rich plasma application — At our pilonidal care clinic, patients will undergo a comprehensive treatment regimen starting with manual or laser hair removal to reduce hair by over 90%. For pilonidal abscesses, we will perform incision, drainage, and antibiotic therapy. Treatments will include local anesthesia with lidocaine and epinephrine, thorough disinfection with povidone-iodine, and wound irrigation. Sinuses will be treated by removing hair and curettage, followed by protective ointment application and crystallized phenol to fill the cavity, ensuring precise dosing and safety.
  For enhanced healing, crystallized phenol + platelet-rich plasma application patients will receive platelet-rich plasma injections to minimize infection risk and promote tissue regeneration, all under strict sterilization to maintain cleanliness and efficacy.
  Arms: Crystallized phenol + platelet rich plasma
Procedure: crystallized phenol — At our pilonidal care clinic, patients will undergo a comprehensive treatment regimen starting with manual or laser hair removal to reduce hair by over 90%. For pilonidal abscesses, we will perform incision, drainage, and antibiotic therapy. Treatments will include local anesthesia with lidocaine and epinephrine, thorough disinfection with povidone-iodine, and wound irrigation. Sinuses will be treated by removing hair and curettage, followed by protective ointment application and crystallized phenol to fill the cavity, ensuring precise dosing and safety.
  Arms: Crystallized phenol

SUMMARY:
The use of local liquid phenol for pilonidal sinus disease was first introduced by Maurica and Greenwood in 1964. Phenol, also known as carbolic acid, has been proven to be an effective sclerosing agent for treating pilonidal sinus diseas. Its antiseptic and anesthetic qualities make it suitable for application in awake patients under local anesthesia. The treatment of pilonidal sinus diseas in children with crystallized phenol was first published by Ateş et al in 2018. However, the treatment involving only crystallized phenol can require numerous sessions, potentially extending the duration of the treatment. IIn this study, the investigators, investigated whether the application of platelet-rich plasma following crystallized phenol treatment could accelerate the healing process and reach better outcomes. This study evaluates the efficacy of PRP as a treatment modality for pilonidal sinus disease in pediatric patients.

DETAILED DESCRIPTION:
Upon their arrival at our pilonidal care clinic, patients commenced a regimen of manual shaving of the gluteal cleft either weekly or bi-weekly. Laser epilation therapy was initiated at the earliest opportunity, conducted every 6 to 8 weeks, aiming for a hair reduction of over 90%. For patients presenting with a pilonidal abscess, an initial procedure of incision and drainage was performed, followed by antibiotic therapy. In the outpatient clinic, patients were placed in a prone position, and the area was sterilized with a povidone-iodine solution.

Anaesthesia local: The skin and subcutaneous tissues surrounding the PSD area, including the sinus openings, receive local anesthesia with 5 ml of lidocaine (20 mg/ml) mixed with epinephrine (0.0125 mg/ml).

Zone keeps clean: The area surrounding the PSD is thoroughly disinfected with povidone-iodine solution, covering a minimum area of 20 square centimeters to ensure adequate local disinfection.

Irrigation with isotonic solution: The wound is washed with sterile isotonic solution.

Zero hair (removing hair and curettage): For sinuses measuring ≤ 3 mm in diameter, dilation is performed using a mosquito clamp (BH-109, Aesculap®, Center Valley, PA, USA). Hair within the sinus is removed. After the complete removal of hair from the area, the granulation tissue is then excised through curettage.

Ointment application around the wound: To prevent skin necrosis and burns, a 0.2% nitrofurazone (Furacin® Eczacıbası İlaç San, Istanbul, Turkey) ointment is meticulously applied around the pilonidal sinus area immediately before the CP application, ensuring a protective barrier and enhancing skin safety.

Gravel-like crystallized phenol application: In this instance, the phenol applied is not in liquid form; rather, it is in a solid, gravel-like form. CP (BotaFarma İlaç Medikal İtriyat Kimya San. Tic. Ltd. Şti, Ankara, Turkey) is carefully administered into the cavity via the orifice, with the precise amount required just sufficient to fill the cavity without causing any overflow. This step necessitates meticulous attention to ensure the correct dosage and prevent any potential spillage. Typically, for an average pediatric patient and the size of the defect encountered, an amount ranging from 4 to 6 grams of phenol is deemed adequate to effectively treat the area while minimizing risk.

Local re-disinfection prior to PRP injection: Up to this point, all procedures are identical for both groups. However, the following steps and any subsequent applications are exclusively for Group 2. The area around the pilonidal sinus should be thoroughly disinfected again with povidone-iodine (care should be taken to prevent povidone-iodine from entering the sinus itself). This step is critical because, following this phase, a PRP injection will be administered into the tissue, necessitating that the skin is properly disinfected to minimize the risk of infection.

Undergo PRP injection: In Group 2, patients received a PRP injection during the same session as the CP application. The amount of PRP injected-approximately 1-2 ml, depending on the size of the pilonidal sinus-was administered around the edges and surrounding area of the wound.

ELIGIBILITY:
Inclusion Criteria:

The study will be included patients with pilonidal sinus disease aged between 0 to 18 years.

Exclusion Criteria:

Patients who had undergone prior pilonidal sinus disease surgery or had anomalies in the sacrococcygeal region will be excluded from the study. Additionally, patients who will decline to participate in the study or will be failed to attend post-procedural outpatient follow-ups will also be excluded.

Ages: 1 Day to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 100 (Estimated)
Dates: Start 2023-11-21 (Actual); Primary Completion 2024-09-29 (Estimated); Study Completion 2024-09-30 (Estimated)

PRIMARY OUTCOMES:
Average time to full daily activities | 1 week
  It refers to the time when patients return to their routine lives after the procedure.
VAS scores | 2 weeks
  Patient visual analog scale (VAS) scores will be assessed both prior to the procedure and again 10 days following the procedure.
Healing time | 7 weeks
  It refers to the wound healing time of the patients after the procedure.
Cosmetic score | 7 weeks
  All patients will be assessed for cosmetic score after healing. For cosmetic evaluation, observers were asked to assess the scar in comparison to normal skin by answering the question, "What is your overall opinion of the scar compared to normal skin?" They rated the scar on a scale from 1 to 10, where 10 signifies normal skin and 1 represents a very different, worst possible scar.
Success rate | 7 weeks
  The succes rate will be calculated after interventions
Recurrence rate | 7 weeks
  The recurrence rate will be calculated after interventions

SECONDARY OUTCOMES:
Bleeding rate | 1 week
  Bleeding during interventions will be calculated
Infection rate | 7 weeks
  Infection will be defined during interventions and 10 days after intervention
Skin burn rate | 7 weeks
  Skin burn during interventions will be calculated
Total complication rate | 7 weeks
  Total complicaitons during interventions will be calculated

CONTACTS AND LOCATIONS:
Locations (1):
- Mustafa Azizoğlu, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Azizoglu M, Klyuev S, Kamci TO, Okur MH. Platelet-rich Plasma as an Adjuvant Therapy to Crystallized Phenol in the Treatment of Pediatric Pilonidal Sinus Disease: A Prospective Randomized Controlled Trial. J Pediatr Surg. 2025 Jan;60(1):161934. doi: 10.1016/j.jpedsurg.2024.161934. Epub 2024 Sep 14. PMID 39307596